CLINICAL TRIAL: NCT00383565
Title: A Phase II Study of Depsipeptide, a Histone Deacetylase Inhibitor, in Relapsed or Refractory Mantle Cell or Diffuse Large Cell Non-Hodgkin's Lymphoma
Brief Title: FR901228 in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00240; NCI-2009-00240 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2005-0579; CDR0000486326; 2005-0579 (Other: M D Anderson Cancer Center); 7869 (Other: CTEP); P30CA016672 (NIH); N01CM62202 (NIH)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — romidepsin

ARMS (1):
- Arm I (Experimental): Patients receive FR901228 IV over 4 hours on days 1, 8, and 15.
  Interventions: Drug: romidepsin

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax

SUMMARY:
FR901228 may stop the growth of cancer cells by blocking some of the enzymes needed for cell to grow and by blocking blood flow to the cancer. This phase II trial is studying how well FR901228 works in treating patients with relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate (complete and partial) to FR901228 in patients with relapsed or refractory mantle cell or diffuse large cell non-Hodgkin's lymphoma.

II. Evaluate the safety and feasibility of FR901228, in terms of the incidence of toxicity and maximum grade observed and courses delayed or dose reductions, in these patients.

III. Determine 2-year progression-free and overall survival.

OUTLINE: Patients receive FR901228 IV over 4 hours on days 1, 8, and 15.

Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed aggressive B-cell non-Hodgkin's lymphoma of 1 of the following subtypes:

  * Mantle cell lymphoma
  * Diffuse large cell lymphoma
  * (Ineligible for or unwilling to undergo stem cell transplantation)
* Relapsed or refractory disease:

  * Any number of prior therapies allowed for relapsed disease, including peripheral blood stem cell or bone marrow transplantation
  * No more than 2 prior regimens, excluding monotherapy with monoclonal antibody or radiotherapy, for refractory disease
* Measurable disease, defined as >= 1 lesion >= 1.5 cm in the longest diameter
* No transformed lymphoma, defined as the transformation of a low-grade lymphoma, including follicular lymphoma or small lymphocytic lymphoma, to a high-grade lymphoma (e.g., diffuse large cell lymphoma)
* ECOG performance status 0-2
* Absolute neutrophil count >= 1,000/mm^3 OR >= 500/mm^3 if extensive bone marrow involvement (> 50%) or hypersplenism with palpable splenomegaly
* Platelet count >= 75,000/mm^3 OR >= 50,000/mm^3 if extensive bone marrow involvement (> 50%) or hypersplenism with palpable splenomegaly
* Bilirubin normal
* Alkaline phosphatase =< 2 times upper limit of normal (ULN)
* AST =< 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant cardiac disease, including New York Heart Association class III-IV congestive heart failure
* No history of serious ventricular arrhythmia
* QTc < 500 msec
* No evidence of cardiac hypertrophy on ECG
* No known HIV positivity
* No other uncontrolled serious medical condition or active infection (e.g., chronic obstructive pulmonary disease, diabetes)
* Recovered from prior therapy
* No prior doxorubicin hydrochloride >= 450 mg/m^2 or mitoxantrone >= 112 mg/m^2 (Patients who received both mitoxantrone and doxorubicin hydrochloride should have a "doxorubicin equivalent dose" < 450 mg/m^2
* No prior therapy with a histone deacetylase inhibitor
* No concurrent dexamethasone or prednisone except for refractory nausea/vomiting
* No concurrent drugs associated with QTc prolongation (e.g., dolasetron mesylate)
* Concurrent hydrochlorothiazide, furosemide, or other diuretics allowed provided patient is receiving potassium chloride supplementation (No supplementation needed if switched to a potassium-conserving diuretic)
* No CNS lymphoma
* Creatinine normal
* Cardiac function >= 50% by MUGA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Romaguera, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 20, 2006 to May 08, 2009. All recruitment done at UT MD Anderson Cancer Center.
Groups:
- FR901228: 13 mg/m^2 FR901228 by vein (IV) over 4 hours on days 1, 8, and 15
Period: Overall Study
Arm/Group | FR901228
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FR901228
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate (Complete Response [CR] and Partial Response [PR]) After 6 Courses of Treatment
Description: International Working Group response for non- Hodgkin's lymphoma: Complete Response (CR) - disappearance all detectable clinical/radiographic evidence of disease and disappearance of all disease-related symptoms (present before therapy) and normalization of those biochemical abnormalities; Partial Response (PR) - ≥50% decrease in sum products of greatest diameters (SPD) of 6 largest dominant nodes or nodal masses, selected by clearly measurable in at least two perpendicular dimensions, from disparate regions of body and no decrease in size of other nodes, liver, or spleen.
Time Frame: 24 weeks (6 courses of 4 week cycles)
Measure: Number; unit: participants
Arm/Group | FR901228
Number analyzed (Participants) | 9
participants
  Complete Response | 0
  Partial Response | 1

2. Secondary Outcome: Median Progression Free-survival (PFS)
Description: Time to disease progression is defined as the time from registration to documentation of disease progression.
Time Frame: 2 Years
Measure: Median (Full Range); unit: months
Arm/Group | FR901228
Number analyzed (Participants) | 9
months | 4 [1 to 7]

3. Secondary Outcome: Median Overall Survival
Description: Survival time is defined as the time from registration to death due to any cause, measured in months. The distribution of survival time estimated using the method of Kaplan-Meier.
Time Frame: 5 Years
Measure: Median (Full Range); unit: months
Arm/Group | FR901228
Number analyzed (Participants) | 9
months | 20 [1 to 53]

ADVERSE EVENTS:
Time Frame: 3 years and 9 months
Arm/Group | FR901228
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FR901228 (N=9)
Neutropenia (Infections and infestations) | 1
Thrombocytopenia (Infections and infestations) | 2
Dysphagia (Gastrointestinal disorders) | 1
Glucose, serum-high (Metabolism and nutrition disorders) | 1
Infection (Infections and infestations) | 1
Diplopia (Eye disorders) | 1
Increased Alkaline phosphatase (Metabolism and nutrition disorders) | 1
Cardiac Arrhythmia (Cardiac disorders) | 1
Death NOS (General disorders) | 1 — NOS = Not Otherwise Specified
Infectious Endocarditis (Cardiac disorders) | 1
Non-neutropenic fever (General disorders) | 1
DVT, Vascular access-related (Vascular disorders) | 1 — Deep vein thrombosis = DVT
Fatigue (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FR901228 (N=9)
weight loss (Investigations) | 2
nausea (Gastrointestinal disorders) | 6
fatigue (General disorders) | 5
thrombocytopenia (Investigations) | 8
anemia (Blood and lymphatic system disorders) | 7
hyperglycemia (Metabolism and nutrition disorders) | 4
anorexia (Metabolism and nutrition disorders) | 2
hypocalcemia (Metabolism and nutrition disorders) | 2
hypoalbuminemia (Metabolism and nutrition disorders) | 4
hyperuricemia (Metabolism and nutrition disorders) | 1
hypoglycemia (Metabolism and nutrition disorders) | 1
hyperkalemia (Metabolism and nutrition disorders) | 4
hypomagnesemia (Metabolism and nutrition disorders) | 2
hyponatremia (Metabolism and nutrition disorders) | 2
blurry vision (Eye disorders) | 2
constipation (Gastrointestinal disorders) | 3
diarrhea (Gastrointestinal disorders) | 3
gastritis (Gastrointestinal disorders) | 1
hemorrhoids (Gastrointestinal disorders) | 1
mucositis oral (Gastrointestinal disorders) | 1
oral pain (Gastrointestinal disorders) | 1
periodontal disease (Gastrointestinal disorders) | 1
rectal pain (Gastrointestinal disorders) | 1
stomach pain (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 3
fever (General disorders) | 2
edema limbs (General disorders) | 2
infection with normal Absolute neutrophil count (ANC) (Infections and infestations) | 7
sinusitis (Infections and infestations) | 1
alanine aminotransferase (ALT) (Investigations) | 2
aspartate aminotransferase (AST) (Investigations) | 3
alkaline phosphatase (Investigations) | 3
creatinine (Investigations) | 1
lymphopenia (Investigations) | 6
leukopenia (Investigations) | 3
neutropenia (Investigations) | 2
hypotension (Vascular disorders) | 1
sensory neuropathy (Nervous system disorders) | 2
dizziness (Nervous system disorders) | 2
myalgia (Musculoskeletal and connective tissue disorders) | 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
sinus tachycardia (Cardiac disorders) | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
taste alteration (Gastrointestinal disorders) | 1
hypophosphatemia (Metabolism and nutrition disorders) | 3
headache (Nervous system disorders) | 1
pruritus (Skin and subcutaneous tissue disorders) | 1
thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less